CLINICAL TRIAL: NCT02636335
Title: Light, Exercise Intensity and Mood in Overweight
Acronym: LEXI-MO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Head of Departement of Sport, Exercise and Health, Principal Investigator, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEXI-MO
Record Dates: First submitted 2015-12-14; First posted 2015-12-21 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Overweight, Obesity Grade I
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright Light (Experimental): 8 a.m. study participants will be exposed to Bright Light (4500 lx) Phillips Energy Light HF3319 for 30 minutes prior and during a 30 minute lasting exercise test with self-chosen exercise intensity on a bicycle ergometer.
  The light exposure and time-trial will be performed in three repetitive exercise sessions 48h apart.
  Interventions: Device: Phillips Energy Light HF3319
- Control (Experimental): 8 a.m. study participants will be exposed to a Control Light Condition (230 lx) Phillips Energy Light HF3319 for 30 minutes prior and during a 30 minute lasting exercise test with self-chosen exercise intensity on a bicycle ergometer.
  The light exposure and time-trial will be performed in three repetitive exercise sessions 48h apart.
  Interventions: Device: Phillips Energy Light HF3319

INTERVENTIONS:
Device: Phillips Energy Light HF3319 — Exposure to Light administered with Phillips Energy Light HF3319.

SUMMARY:
The purpose of this study is to determine if an exposure to light in the morning has a positive influence on self-chosen exercise intensity on a bicycle ergometer in overweight and obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 25 - 35 kg/m2

Exclusion Criteria:

* Women who are pregnant or breast feeding,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Participation in other studies in the last four weeks
* Systolic blood pressure > 170 mmHg, diastolic blood pressure > 100 mmHg
* Shift work in the last two months
* Travels across time zones in the last four weeks
* Use of photosensitisation drugs
* Clinical manifest depression
* Cardiovascular diseases which reduce age-appropriate exercise capacity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Mean power output in watts | Power output during the first 30 minute time-trial on a bicycle ergometer.

SECONDARY OUTCOMES:
Subjective sleepiness | 1 minute after the light exposure vs. 1 minute before the light exposure in the first time trial
  Subjective sleepiness will be measured with the Multidimensional Mood Questionnaire (Category "Wakefulness - Sleepiness")
Subjective Mood | 1 minute after the light exposure vs. 1 minute before the light exposure in the first time trial
  Subjective Mood measured with the Multidimensional Mood Questionnaire (Category "Good Mood - Bad Mood")
Mean power output in watts during the first, second and third time-trial on a bicycle ergometer. | Mean of the 30 minutes of the exercise from the first, second and third time-trial.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof., Principal Investigator — University of Basel
Locations (1):
- Departement of Sport, Exercise and Health, Basel, Switzerland